CLINICAL TRIAL: NCT04499183
Title: A Feasibility Study on Fiber Fermentation, and Short Chain Fatty Acid Kinetics and Utilization Inside the Gut and Systemic Circulation
Brief Title: Fiber Fermentation, and Short Chain Fatty Acid Kinetics and Utilization Inside the Gut and Systemic Circulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NL74418.081.20
Record Dates: First submitted 2020-02-26; First posted 2020-08-05 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-digestible carbohydrates (Experimental): fructo- and galacto-oligosaccharides
  Interventions: Dietary Supplement: fructo- and galacto-oligosaccharides
- placebo (Placebo Comparator): maltodextrin
  Interventions: Dietary Supplement: fructo- and galacto-oligosaccharides

INTERVENTIONS:
Dietary Supplement: fructo- and galacto-oligosaccharides — 15 gram/day fructo- and galacto-oligosaccharides
  Other Names: FOS and GOS

SUMMARY:
Nowadays there is a strong interest in optimising human health through manipulation of non-digestible carbohydrates (NDC). NDC can be used as substrates by gut microbiota, which results in NDC degradation, production of fermentation products, such as short-chain fatty acids (SCFA), and a shift in microbiome composition and activity. It is hypothesized that SCFAs mediate parts of the beneficial effects of NDC. In mice, the influx of SCFA into the host correlated strongly with improvements of markers of the metabolic syndrome, in contrast to the concentrations of SCFA in the proximal colon. Therefore, the influx of short chain fatty acids (SCFA) into the body may be of high importance in improving metabolism. There is a need for more studies in humans to trace the life course of SCFA and their regulatory role in human metabolism. To study this inner world of bacterial products in humans, we will use a nasal-intestine catheter that can be used for delivery of components and sampling chyme in the proximal colon. Before the proposed methodology can be applied in a large intervention study, a small scale feasibility study needs to be performed that addresses colonic placement of the nasal-intestine cathether and colonic sampling of regular and NDC-enriched chyme samples. We will investigate the acute fermentation of fructo- and galacto-oligosaccharides in the proximal colon. Moreover, we will deliver 13C-labelled SCFA via a naso-intestinal catheter to quantify the fluxes of SCFA production, interconversion and uptake by the host. A small-scale, 7-day parallel feasibility trial, N=5 subjects will receive GOS/FOS supplements (mix 1:1 ratio, 15 gram/day), and N=5 other subjects will receive placebo supplements (isocaloric maltodextrin, 12 gram/day). At the last day of the supplementation period, the catheter will be placed, and afterwards participants stay maximum 5 hours in the hospital, to ensure progression of the nose-intestine catheter. After an overnight fast, subjects will visit the hospital again for measurements. Subjects will consume a NDC bolus (200 mL tap water, 5 gram fructo-oligosaccharides, 5 gram galacto-oligosaccharides, non-absorbable marker (PEG-4000). Afterwards, they are not allowed to eat for 6.5 hours. Isotopically 13C-labelled SCFAs will be delivered in the proximal colon. Blood and colonic luminal samples, breath samples, faeces and urine will be collected.

ELIGIBILITY:
Inclusion criteria:

* Males
* Age 18-60yrs
* BMI between 18.5 and 30 kg/m2
* Regular bowel movement (defaecation on average once a day)
* Signed informed consent

Exclusion criteria:

* Having a history of medical or surgical events that, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results of the study (e.g. diabetes, cardiovascular disease, gastrointestinal disease, renal failure, cancer, infectious disease, nose/throat).
* Having a history of surgical events of the gastro-intestinal tract (e.g. bariatric surgery/gastric bypass surgery)
* Presence of swallowing disorder
* Use of any prescribed or non-prescribed medication (other than paracetamol) including antacids, analgesics, and herbal remedies during the three (3) weeks prior to study start.
* Being lactose intolerant
* Follows a vegan diet
* Use of antibiotics within 3 months of starting the study or planned during the study
* Use of pro- or prebiotics (e.g. galacto-oligosaccharides, fructo-oligosaccharides)
* Constipation/infrequent bowel movement (less than 3 times defaecation per week)
* Abuse of drugs/alcohol (alcohol: >4 consumptions/day or >21 consumptions/week)
* Smoker
* Having diarrhoea within 1 month prior to the study start
* Personnel of Wageningen University, Division of Human Nutrition, their partner and their first and second degree relatives
* Participation in another biomedical study or other research from the Division of Human Nutrition
* Not willing to be exposed to fluoroscopy
* Having a hemoglobin of <8.5 mmol/L
* Having blood vessels that are too difficult for inserting a cannula
* Not having a general practitioner

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Concentrations of carbohydrates | Between 0 and 400 minutes
  mono-, di-, tri-, oligo- and polysaccharides in the intestinal lumen
Relative microbiota composition and metabolites | Between 0 and 400 minutes
  Microbiota and metabolites inside the intestine
Concentrations of plasma metabolites | Between 0 and 400 minutes
  organic acids, amino acids, glucose, cholesterol, fatty acids and bile acids in blood
Catheter placement in the colon | After 1 week
  To show placement of a naso-intestinal catheter in the proximal colon.
Volume of colon sample (mL) | Between 0 and 400 minutes
  To check whether enough material for analysis is obtained if the catheter system takes samples in the proximal colon of participants.
Concentrations of SCFAs | Between 0 and 400 minutes
  (13C isotopic) enrichments of SCFAs inside intestinal lumen

SECONDARY OUTCOMES:
Concentrations of urine metabolites | After 0 and 120 minutes
  hippurate, di- en tri-methylamine, acetaldehydes, taurine, glycine, glucuronic acid conjugates, and bile acid profiles (conjugates)
Questionnaires about (dis)comfort of study procedures | After 1 week
  Questions about study procedures
Relative microbiota composition and metabolite concentrations | After 1 week
  Microbiota and metabolome in faeces

OTHER OUTCOMES:
Concentrations of non-digestible markers | Between 0 and 400 minutes
  TiO2 and PEG-4000 inside the intestine

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University and Research, Wageningen, Netherlands